CLINICAL TRIAL: NCT06356857
Title: Assessing Repeatability and Intra-individual Variability in [O15]H2O-PET Myocardial Perfusion Imaging
Acronym: Heart-Wave
Status: Active, not recruiting | Type: Observational
Sponsor: Peter Hovind (Other)
Responsible Party: Sponsor-Investigator, Peter Hovind, Head of department, Department of Clinical Physiology and Nuclear Medicine and PET, Bispebjerg Hospital
Organization: Bispebjerg Hospital (Other)
Other Study IDs: H-23070312
Record Dates: First submitted 2024-03-13; First posted 2024-04-10 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2024-08

CONDITIONS: Myocardial Blood Flow
MeSH Terms: interventions — Myocardial Perfusion Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- re-pet participant: Participant are enrolled for a second pet-scan which will be compared with the initial scan.
  Interventions: Diagnostic Test: Myocardial perfusion imaging (MPI) using [O15]H2O-PET-CT

INTERVENTIONS:
Diagnostic Test: Myocardial perfusion imaging (MPI) using [O15]H2O-PET-CT — Re-scan for comparison with initial scan

SUMMARY:
This study wish to assess the reproducibility of baseline and hyperemic myocardial blood flow as well as myocardial blood flow reserve measurements with [O15]H2O-PET-MPI.

DETAILED DESCRIPTION:
Myocardial perfusion imaging (MPI) using [O15]H2O-PET-CT represents a validated technique for quantitatively assessing myocardial blood flow (MBF) and myocardial flow reserve (MFR).

With advancements in scanner and software technology, it is now possible to accurately quantify both global and regional MBF in clinical PET-MPI studies. Reduced stress MBF or MFR, as determined by [O15]H2O-PET-MPI, is a reliable indicator for detecting hemodynamically significant coronary artery stenosis. Additionally, MBF and MFR offer valuable prognostic insights into mortality and the risk of myocardial infarction. Clinical experience suggests that implementing [O15]H2O-PET-MPI for coronary artery disease evaluation is not only feasible but also aids in making informed decisions regarding revascularization.

This study wish to assess the reproducibility of baseline and hyperemic myocardial blood flow as well as myocardial blood flow reserve measurements with [O15]H2O-PET-MPI.

ELIGIBILITY:
Inclusion Criteria:

* Patients > 50 years of age referred for [O15]H2O-PET-MPI by the dept. of cardiology on clinical indication with symptoms suggestive of myocardial ischemia, primarily angina.
* Willing to repeat the [O15]H2O-PET-MPI
* Normal left ventricular ejection fraction (EF > 45), as assessed from recent (max 1 year old) echocardiography description in medical journal.

Exclusion Criteria:

* Cardiovascular event in between scans (defined as hospitalization for cardiovascular event).
* History of myocardial infarction
* Regional perfusion deficits on the primary [O15]H2O-PET-MPI clinically suspected as a sign of significant coronary stenosis.
* Unstable angina
* Severe Chronic Obstructive Pulmonary Disease (COPD)
* Severe asthma
* Claustrophobia
* Acute illness
* Significant language barrier, estimated by the investigator not being able to understand the study information sufficiently.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients > 50 years of age with symptoms suggestive of myocardial ischemia, primarily angina. They have therefore undergone [O15]H2O-PET-MPI by the dept. of cardiology on clinical indication.
  The investigators will include 50% women.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-15 (Actual); Primary Completion 2025-03-17 (Actual); Study Completion 2026-03-17 (Estimated)

PRIMARY OUTCOMES:
[O15]H2O-PET-MPI variability and repeatability coefficient estimated from 20 patients having [O15]H2O-PET-MPI done twice | 8 months
  In this study two [O15]H2O-PET-CT scans in the same induvidual at two different timepoints will be conducted. This will allow a variability estimation (for each meassurement eg rest MBF (ml/g/min), stress MBF (ml/g/min)) and thereby a calculated repeatability coefficient.

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hovind, MD, Phd., Study Chair — Bispebjerg hospital, capitol region Denmark
Locations (1):
- Bispebjerg Hospital, Copenhagen, RegionH, Denmark

IPD SHARING:
Plan to Share IPD: No